CLINICAL TRIAL: NCT03180632
Title: Effect of A Single Dose of Lorazepam on Salivary Cortisol Response in Children Undergoing Digestive Endoscopy: a Randomized Double Blinded Study
Brief Title: Effect of A Single Dose of Lorazepam on Salivary Cortisol Response in Children Undergoing Digestive Endoscopy:
Acronym: Endo-Lora
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: St. Justine's Hospital (Other)
Responsible Party: Principal Investigator, Jantchou Prevost, MD,PhD, St. Justine's Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: JP2017
Record Dates: First submitted 2017-06-02; First posted 2017-06-08 (Actual); Last update posted 2018-09-05 (Actual); Status verified 2018-09

CONDITIONS: Anxiety
MeSH Terms: conditions — Anxiety Disorders | interventions — Lorazepam

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Group A (Active Comparator): Patient will receive a single dose of either 0,5mg or 1mg of oral Lorazepam depending on their body weight.
  Interventions: Drug: Lorazepam
- Group B (Placebo Comparator): Patient will receive a placebo similar in color, form and size.
  Interventions: Other: Placebo
- Group 3 (No Intervention): Patient will receive no intervention.

INTERVENTIONS:
Drug: Lorazepam — Patient receives one or two tablet of 0,5mg Lorazepam according to body weight
  Other Names: Apo-Lorazepam
  Arms: Group A
Other: Placebo — Patient receive one of two tablet of Placebo according to body weight
  Arms: Group B

SUMMARY:
The purpose of this study is to determine the effect of a single dose of Lorazepam on salivary cortisol in children undergoing digestive endoscopy. To do so, the patients will be randomized in three groups. The first group receives the Lorazepam, the second group receives a placebo and the last group receives no intervention. Each patient will have three saliva samples taken at three different time point on the day of the endoscopy and will be asked to fill out questionnaires on anxiety and overall satisfaction of the procedure.

DETAILED DESCRIPTION:
Background: Pediatric digestive endoscopies (gastroscopy and colonoscopy) are invasive procedures. All endoscopic procedure are conducted in the operating room either under intravenous (IV) sedation or general anesthesia. More than 50% of procedures are performed using IV sedation. The current sedation protocol in the endoscopy suite is a combination of Midazolam (0.1 mg/kg) and Fentanyl (1 microgram/kg) in all children. The children undergoing colonoscopies receive and additional administration of Ketamine (0.5 mg/kg).

In a previous study performed in children 10-18 years undergoing upper and lower endoscopy, the investigators found that despite this regimen, 25% of the children expressed a significantly high level of pain during endoscopy under IV sedation.

Because general anesthesia is not available for all children, it is important to investigate strategies that could help in minimizing the discomfort and pain during the procedure.

Salivary cortisol (sCortisol) has been used in several pediatric studies to determine the level of stress in children prior to various medical procedures. In another study done at our site, the investigators have found sCortisol to be a reliable biomarker of stress for children undergoing digestive endoscopies. Furthermore, the mean baseline sCortisol levels were higher in the group that experienced procedural pain.

Lorazepam is a a rapid onset benzodiazepine that has anxiolytic and sedative properties that has been approved by Health Canada as an adjunct therapy for the relief of excessive anxiety that might be present prior to surgical interventions.

Objective:

The primary objective is to investigate the effect of Lorazepam as compared to placebo on the change of the level of sCortisol between baseline (C1) and immediately before endoscopy (C2) in adolescents undergoing a gastroscopy or a colonoscopy. The investigators think that it might be possible to modulate the stress response with the administration of a benzodiazepine as soon as the children arrives at the hospital. Thus children could have a better experience of the digestive endoscopic procedure (less pain and more comfort).

The secondary outcome measure will be:

(1) the proportion of children experiencing procedural pain, (2) the duration of endoscopic procedures, (3) children satisfaction, (4) physician and nurse satisfaction (5) the total dose of Fentanyl and Ketamine per kilogram body weight delivered during the procedure and (6) the mean change between pre-op and postop cortisol levels between the two groups.

Safety outcomes measures: The following adverse events will be sought before and during the endoscopy: prolonged drowsiness, hypotension, hypertension, desaturation, bradycardia.

Exploratory outcomes: the mean change between pre-op and postop cortisol levels in the Group C (No intervention) compared to Group A and B.

Methods:

In this randomized controlled trial children will be assigned to one of the three following groups (no intervention, placebo and active drug). The investigators will collect salivary samples to measure the levels of sCortisol and investigate their variation between three timepoint ( at arrival at the hospital, right before the procedure and right after the procedure). sCortisol levels will be correlated to a questionnaire evaluating the anxiety level in the patient. The research team will also evaluate the pain experienced during the procedure using the Nurse-Assessed Patient Comfort Score (NAPCOMS): a validated tool for the evaluation of pain in subjects undergoing endoscopies).

ELIGIBILITY:
Inclusion Criteria:

* Children aged 9-18 seen in our endoscopic unit
* Children undergoing upper, lower or combined digestive endoscopy
* Procedure to be performed within 3 hours of inclusion in the study and drug administration

Exclusion Criteria:

* Unable to read or speak English or French
* Diagnosed with a psychiatric or neurological disorder
* Myasthenia gravis
* Acute narrow angle glaucoma
* Known hypersensitivity to benzodiazepines
* Already treated with an anxiolytic on a regular basis
* Receiving a drug contraindicated in association with benzodiazepines
* Receiving oral, intravenous or inhaled corticosteroids in the last two days before randomization
* Body weight less than 20 kg
* Pregnancy

Ages: 9 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 98 (Actual)
Dates: Start 2017-06-28 (Actual); Primary Completion 2018-06-01 (Actual); Study Completion 2018-06-01 (Actual)

PRIMARY OUTCOMES:
Change of sCortisol from baseline to one hour after drug administration | One hour after drug administration
  Proportion of children with a decrease of sCortisol of at least 15 points between the group Placebo and the group Lorazepam

SECONDARY OUTCOMES:
Procedural pain | during endoscopic procedure
  Proportion of children experiencing procedural pain
Duration of endoscopic procedure | Through completion of endoscopy: an average of 2 hours after drug administration
  Duration of endoscopic procedure. The time interval in minutes will be measured between the start and the end of each procedure.
Children Satisfaction | Through study completion, an average of 3 hours
  Children satisfaction will be evaluated with a validated Satisfaction questionnaire of children undergoing endoscopy
Physician Satisfaction | during the endoscopic procedure
  Physician satisfaction will be evaluated with a validated tool : CLINICIAN SATISFACTION WITH SEDATION INSTRUMENT (CSSI)
Nurse Satisfaction | during the endoscopic procedure
  Nurse satisfaction will be evaluated with a validated tool : NURSE ASSESSED PATIENT COMFORT SCORE (NAPCOMS)
Medication needed For sedation | during the procedure
  Total dose of Fentanyl and Ketamine per kilogram body weight delivered
Change in sCortisol levels between pre-op and post-op | one hour after the endoscopic procedure
  Mean change between pre-op and post-op cortisol levels between the two groups (Lorazepam and Placebo)

OTHER OUTCOMES:
Number of participants with Treatment-related Adverse Events (Safety and Tolerability) | during the procedure
  The following adverse events will be sought before and during the endoscopy: prolonged drowsiness, hypotension, hypertension, desaturation, bradycardia.
Change in level of sCortisol between pre-op and post-op in the group without any intervention | Through study completion, an average of 3 hours
  the mean change between pre-op and post-op cortisol levels in the Group C (No intervention)

CONTACTS AND LOCATIONS:
Overall Officials: Prévost Jantchou, MD, PhD, Principal Investigator — Ste-Justine Hospital
Locations (1):
- CHU Sainte-Justine, Montreal, Quebec, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Chennou F, Bonneau-Fortin A, Portolese O, Belmesk L, Jean-Pierre M, Cote G, Dirks MH, Jantchou P. Oral Lorazepam is not Superior to Placebo for Lowering Stress in Children Before Digestive Endoscopy: A Double-Blind, Randomized, Controlled Trial. Paediatr Drugs. 2019 Oct;21(5):379-387. doi: 10.1007/s40272-019-00351-9. PMID 31418168